CLINICAL TRIAL: NCT02166476
Title: Phase III, Randomized, Double-Blind, Study Evaluating Efficacy/Safety/Tolerability of Meropenem-Vaborbactam Compared to Piperacillin/Tazobactam in Adult Patients With Complicated Urinary Tract Infections, Including Acute Pyelonephritis
Brief Title: Efficacy/Safety of Meropenem-Vaborbactam Compared to Piperacillin-Tazobactam in Adults With cUTI and AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rempex 505
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-04

CONDITIONS: Urinary Tract Infection Complicated; Acute Pyelonephritis
MeSH Terms: interventions — meropenem and vaborbactam; Meropenem; beta-Lactamase Inhibitors; vaborbactam; Piperacillin, Tazobactam Drug Combination; Piperacillin; Tazobactam; Levofloxacin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind-double dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meropenem-Vaborbactam (Experimental): Meropenem-vaborbactam (meropenem 2 grams [g] plus vaborbactam 2 g), infused in 250 milliliters (mL) normal saline, administered intravenously (IV) over 3 hours, every 8 hours (q8h), with 100 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-milligram (mg) dose every 24 hours (q24h) after a minimum of 15 doses of IV meropenem-vaborbactam plus saline, if clinically indicated. Total treatment was 10 days, unless a participant had baseline bacteremia where up to 14 days of therapy could be administered IV.
  Interventions: Drug: Meropenem-Vaborbactam; Drug: Levofloxacin; Drug: Saline
- Piperacillin-Tazobactam (Active Comparator): Piperacillin-tazobactam (piperacillin 4 g plus tazobactam 0.5 g), infused in 100 mL normal saline, administered IV over 30 minutes, q8h, with 250 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after a minimum of 15 doses of IV piperacillin-tazobactam plus saline, if clinically indicated. Total treatment was 10 days, unless a participant had baseline bacteremia where up to 14 days of therapy could be administered IV.
  Interventions: Drug: Piperacillin-Tazobactam; Drug: Levofloxacin; Drug: Saline

INTERVENTIONS:
Drug: Meropenem-Vaborbactam — Meropenem-vaborbactam
  Other Names: Combination vaborbactam and meropenem; beta-lactamase inhibitor and carbapenem antibiotic; Carbavance; Vabomere; Meropenem 2 g-Vaborbactam 2 g
  Arms: Meropenem-Vaborbactam
Drug: Piperacillin-Tazobactam — Piperacillin-tazobactam
  Other Names: Piperacillin 4 g-Tazobactam 0.5 g
  Arms: Piperacillin-Tazobactam
Drug: Levofloxacin — Levofloxacin
  Other Names: Levo
Drug: Saline — Saline

SUMMARY:
Meropenem-vaborbactam is being compared to piperacillin-tazobactam in the treatment of adults with complicated urinary tract infection (cUTI) or acute pyelonephritis (AP).

DETAILED DESCRIPTION:
In the current era of increased resistance to extended spectrum cephalosporins, carbapenem antimicrobial agents are frequently the antibiotics of "last defense" for the most resistant pathogens in serious infections, including those found in cUTIs. The recent dissemination of serine carbapenemases in Enterobacteriaceae in many hospitals worldwide now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing meropenem-vaborbactam administered as a fixed combination by intravenous infusion to treat serious Gram-negative infections such as cUTIs, including those infections caused by bacteria resistant to currently available carbapenems.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form, the ability to understand the study conduct and tasks that are required for study participation, and a willingness to cooperate with all tasks, tests, and examinations as required by the protocol.
2. Male or female ≥18 years of age.
3. Weight ≤185 kilograms (kg).
4. Expectation, in the judgment of the Investigator, that the participant's cUTI or AP requires initial treatment with at least 5 days of IV antibiotics.
5. Documented or suspected cUTI or AP as defined below:

   cUTI

   Signs or symptoms evidenced by at least 2 of the following:
   * Chills, rigors, or fever (fever must be documented within 24 hours of the screening visit with a temperature of ≥38.0 degrees Celsius [°C] [≥100.4 degrees Fahrenheit (°F)] or rectal/core temperature ≥38.3°C [≥100.9°F], observed and documented by a health care provider);
   * Elevated white blood cell count (>10,000/ cubic millimeters [mm^3]) or left shift (>15% immature polymorphonuclear leukocytes [PMNs]);
   * Nausea or vomiting;
   * Dysuria, increased urinary frequency, or urinary urgency;
   * Lower abdominal pain or pelvic pain

   Pyuria evidenced by 1 of the following:
   * Positive leukocyte esterase (LCE) on urinalysis;
   * White blood cell count ≥10 cells/mm^3 in unspun urine;
   * White blood cell count ≥10 cells/high-power field (hpf) in urine sediment

   At least 1 of the following associated risks:
   * Indwelling urinary catheter;
   * Neurogenic bladder with presence or history of urine residual volume of ≥100 mL;
   * Obstructive uropathy (such as, nephrolithiasis, tumor, fibrosis) that is expected to be medically or surgically treated within 48 hours post randomization;
   * Azotemia due to intrinsic renal disease;
   * Urinary retention in men due to previously diagnosed benign prostatic hypertrophy

   AP

   Signs or symptoms evidenced by at least 2 of the following:
   * Chills, rigors, or fever (fever must be documented within 24 hours of the screening visit with a temperature of ≥38.0°C [≥100.4°F] or rectal/core temperature ≥38.3°C [≥100.9°F], observed and documented by a health care provider);
   * Elevated white blood cell count (>10,000/mm^3), or left shift (>15% immature PMNs);
   * Nausea or vomiting;
   * Dysuria, increased urinary frequency, or urinary urgency;
   * Flank pain;
   * Costo-vertebral angle tenderness on physical examination

   Pyuria evidenced by 1 of the following:
   * Positive LCE on urinalysis;
   * White blood cell count ≥10 cells/mm^3 in unspun urine;
   * White blood cell count ≥10 cells/hpf in urine sediment
6. Expectation, in the judgment of the Investigator, that any indwelling urinary catheter or instrumentation (including nephrostomy tubes and/or indwelling stents) will be removed or replaced (if removal is not clinically acceptable) before or as soon as possible, but not longer than 12 hours, after randomization.
7. Expectation, in the judgment of the Investigator that the participant will survive with effective antibiotic therapy and appropriate supportive care for the anticipated duration of the study.
8. Women of childbearing potential must have a negative pregnancy test before randomization and be willing to use a highly effective method of contraception between randomization and for 7 days after the completion of the study. A highly effective method of contraception includes 2 of the following: hormonal implants/patch, injectable hormones, oral hormonal contraceptives, prior bilateral oophorectomy, prior hysterectomy, prior bilateral tubal ligation, intra-uterine device, approved cervical ring, condom, true abstinence (if approved by the Investigator), or a vasectomized partner.
9. Willingness to comply with all the study procedures, whether in the hospital or after discharge, for the duration of the study.

Exclusion Criteria:

1. Presence of any of the following conditions:

   1. Perinephric abscess;
   2. Renal corticomedullary abscess;
   3. Uncomplicated urinary tract infection;
   4. Polycystic kidney disease;
   5. Chronic vesicoureteral reflux;
   6. Previous or planned renal transplantation;
   7. Participants receiving hemodialysis;
   8. Previous or planned cystectomy or ileal loop surgery; or
   9. Known candiduria.
2. Presence of suspected or confirmed acute bacterial prostatitis, orchitis, epididymitis, or chronic bacterial prostatitis as determined by history and/or physical examination.
3. Gross hematuria requiring intervention other than administration of study drug.
4. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period (except surgery required to relieve an obstruction or place a stent or nephrostomy).
5. Renal function at screening as estimated by creatinine clearance <50 mL/minute (min) using the Cockcroft-Gault formula.
6. Known non-renal source of infection such as endocarditis, osteomyelitis, abscess, meningitis, or pneumonia diagnosed within 7 days prior to randomization.
7. Any of the following signs of severe sepsis:

   1. Shock or profound hypotension defined as systolic blood pressure <90 millimeters mercury (mmHg) or a decrease of >40 mmHg from baseline (if known) that is not responsive to fluid challenge;
   2. Hypothermia (temperature <35.6°C or <96.1°F); or
   3. Disseminated intravascular coagulation as evidenced by prothrombin time or partial thromboplastin time ≥2 × the upper limit of normal (ULN) or platelets <50% of the lower limit of normal.
8. Pregnant or breastfeeding women.
9. History of epilepsy or known seizure disorder requiring current treatment with anti-seizure medication.
10. Treatment within 30 days prior to enrollment with valproic acid.
11. Treatment within 30 days prior to enrollment with probenecid.
12. Treatment within 30 days prior to enrollment with any cancer chemotherapy, immunosuppressive medications for transplantation, or medications for rejection of transplantation.
13. Evidence of significant hepatic disease or dysfunction, including known acute viral hepatitis or hepatic encephalopathy.
14. Aspartate aminotransferase or alanine aminotransferase >5 × ULN or total bilirubin >3 × ULN.
15. Receipt of any potentially therapeutic antibiotic agent within 48 hours before randomization. Participants with a pathogen-causing cUTI or AP that is resistant to the prior therapy may be enrolled in this study (assuming the organism is known to be sensitive to piperacillin/tazobactam). Participants who develop signs and symptoms of cUTI or AP while on antibiotics may also be enrolled.
16. Prior exposure to vaborbactam alone or in combination with another product.
17. Receipt of any potentially therapeutic antibiotic agent within 48 hours before randomization.

    EXCEPTIONS:
    * Participants who received a single dose of a short-acting oral or IV antibiotic (an antibiotic that is typically dosed every 4 hours, every 6 hours, or q8h in a participant with normal renal function). No more than 25% of participants will be enrolled who meet this criterion.
    * Participants who received >48 hours of prior systemic antibiotic therapy for the current episode of cUTI with unequivocal clinical evidence of treatment failure (that is, worsening signs and symptoms).
    * Participants who develop signs and symptoms of cUTI or AP while on antibiotics for another indication.
18. Requirement at time of enrollment for any reason for additional systemic antibiotic therapy (other than study drug) or antifungal therapy. Topical antifungal or a single oral dose of any antifungal treatment for vaginal candidiasis will be allowed.
19. Likely to require the use of an antibiotic for cUTI prophylaxis during the participant's participation in the study (from enrollment through the last follow up visit).
20. Known history of human immunodeficiency virus infection and known recent cluster of differentiation 4 count <200/mm^3.
21. Presence of immunodeficiency or an immunocompromised condition including hematologic malignancy, bone marrow transplant, or receiving immunosuppressive therapy such as cancer chemotherapy, medications for the rejection of transplantation, and long-term (≥2 weeks) use of systemic corticosteroids.
22. Presence of neutropenia (<1,000 PMNs/mm^3).
23. Presence of thrombocytopenia (<60,000 platelets/mm^3).
24. A corrected QT with Fridericia's Formula >480 milliseconds.
25. History of significant hypersensitivity or allergic reaction to meropenem/vaborbactam, piperacillin/tazobactam, any of the excipients used in the respective formulations, or any beta-lactam antibiotics (such as, cephalosporins, penicillins, carbapenems, or monobactams).
26. Known hypersensitivity or inability to tolerate all of the following: fluoroquinolones (including levofloxacin), trimethoprim/ sulfamethoxazole, cefdinir, cefixime, or cefpodoxime, based on prescribing information.
27. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol.
28. An employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employee or the Investigator.
29. Acute Physiology and Chronic Health Evaluation II score >30 (if clinically indicated)
30. Inability to tolerate intravenous fluids, due to medical reasons, of 1050 mL per day required for study drug administration.
31. Any recent history of trauma to the pelvis or urinary tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fusaro, Study Director — Sponsor GmbH; Keith Kaye, Principal Investigator — Wayne State University
Locations (70):
- United States (8):
  - Mobile, Alabama
  - San Diego, California
  - Denver, Colorado
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - New Brunswick, New Jersey
  - Buffalo, New York
- Belarus (5):
  - Brest
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Brazil (5):
  - São José do Rio Preto, São Paulo
  - Belo Horizonte
  - Campinas
  - Rio de Janeiro
  - São Paulo
- Bulgaria (5):
  - Lovech
  - Montana
  - Silistra
  - Sofia
  - Varna
- Czechia (5):
  - Hradec Králové
  - Karlovy Vary
  - Opava
  - Ústí nad Labem
  - Zlín
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (4):
  - Baja
  - Budapest
  - Debrecen
  - Sopron
- Italy (5):
  - Bologna
  - Catania
  - Florence
  - Perugia
  - Torino
- Peru (5):
  - Arequipa
  - Cusco
  - Ica
  - Lima
  - San Martín de Porres
- Poland (5):
  - Częstochowa
  - Gdansk
  - Kutno
  - Piaseczno
  - Warsaw
- Romania (2):
  - Bucharest
  - Craiova
- Slovakia (4):
  - Poprad
  - Ružomberok
  - Trnava
  - Žilina
- Slovenia (2):
  - Golnik
  - Ljubljana
- Gyeonggi-do, South Korea
- Spain (2):
  - Barcelona
  - Madrid
- Taiwan (2):
  - Kaohsiung City
  - Taichung
- Ukraine (8):
  - Chernivtsi
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Odesa
  - Poltava
  - Vinnitsa
  - Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaye KS, Bhowmick T, Metallidis S, Bleasdale SC, Sagan OS, Stus V, Vazquez J, Zaitsev V, Bidair M, Chorvat E, Dragoescu PO, Fedosiuk E, Horcajada JP, Murta C, Sarychev Y, Stoev V, Morgan E, Fusaro K, Griffith D, Lomovskaya O, Alexander EL, Loutit J, Dudley MN, Giamarellos-Bourboulis EJ. Effect of Meropenem-Vaborbactam vs Piperacillin-Tazobactam on Clinical Cure or Improvement and Microbial Eradication in Complicated Urinary Tract Infection: The TANGO I Randomized Clinical Trial. JAMA. 2018 Feb 27;319(8):788-799. doi: 10.1001/jama.2018.0438. PMID 29486041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Started (5 participants were randomized but not dosed: 4 withdrew consent, 1 did not meet inclusion criteria.) | 272 | 273
Received at Least 1 Dose of Study Drug (Randomized participants included in the Safety and modified intent-to-treat [MITT] populations.) | 272 | 273
Completed | 258 | 250
Not Completed | 14 | 23
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 5 | 10
Not completed — Physician Decision | 1 | 0
Not completed — Unable to Come for Visit | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug (MITT population).
Groups:
- Meropenem-Vaborbactam: Meropenem-vaborbactam (meropenem 2 g plus vaborbactam 2 g), infused in 250 mL normal saline, administered IV over 3 hours, q8h, with 100 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after a minimum of 15 doses of IV meropenem-vaborbactam plus saline, if clinically indicated. Total treatment was 10 days, unless a participant had baseline bacteremia where up to 14 days of therapy could be administered IV.
- Total: Total of all reporting groups
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam | Total
Number analyzed (Participants) | 272 | 273 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (19.42) | 52.6 (20.93) | 52.8 (20.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 180 | 361
  Male | 91 | 93 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 19 | 43
  Not Hispanic or Latino | 248 | 254 | 502
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 254 | 252 | 506
  More than one race | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of Participants In The Microbiological Modified Intent-To-Treat (m-MITT) Population Who Achieved Overall Success At The End Of Intravenous Treatment Visit
Description: This was the primary outcome measure for the Food and Drug Administration (FDA). For this composite outcome measure, overall success was achieved with a clinical outcome of Cure or Improvement and microbiologic outcome of Eradication at the end of intravenous treatment (EOIVT). Cure was defined as the complete resolution or significant improvement of the baseline signs and symptoms. Improvement was defined as lessening, incomplete resolution, or no worsening of the baseline signs and symptoms. Eradication was defined using the FDA's colony-forming units (CFU)/mL criteria that the bacterial pathogen(s) found at baseline was/were reduced to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: EOIVT (Days 5-14)
Population: The m-MITT population included all participants who were randomized, received at least 1 dose of study drug, and had a baseline bacterial pathogen(s) of ≥10^5 CFU/mL of urine at baseline urine culture or the same bacterial pathogen present in concurrent blood and urine cultures.
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem-Vaborbactam: Meropenem-vaborbactam (meropenem 2 g plus vaborbactam 2 g), infused in 250 mL normal saline, administered IV over 3 hours, q8h, with 100 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after a minimum of 15 doses of IV meropenem-vaborbactam plus saline, if clinically indicated. Treatment was administered for up to 14 days.
- Piperacillin-Tazobactam: Piperacillin-tazobactam (piperacillin 4 g plus tazobactam 0.5 g), infused in 100 mL normal saline, administered IV over 30 minutes, q8h, with 250 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after a minimum of 15 doses of IV piperacillin-tazobactam plus saline, if clinically indicated. Treatment was administered for up to 14 days.
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants | 189 | 171
Statistical Analysis 1: Comparison: Meropenem-Vaborbactam vs Piperacillin-Tazobactam; Treatment comparison of the m-MITT population; Test type: Non-Inferiority or Equivalence — The noninferiority margin was a difference of 15%. Noninferiority was concluded if the lower limit of the two-sided 95% confidence interval (CI) for the treatment difference for overall success at EOIVT was >-15%; Treatment difference = 4.5, 95% CI 2-sided [0.7 to 9.1] — Treatment difference is the estimate of the difference in the overall success rate between the two treatment arms. The difference estimates and the 95% CIs are obtained based on Miettinen and Nurminen method

2. Primary Outcome: Proportion Of Participants In The m-MITT Population Who Achieved A Microbiologic Outcome Of Eradication At The Test Of Cure Visit
Description: This was the primary outcome measure for the European Medicines Agency (EMA). For this measure, a microbiologic outcome of Eradication was defined using the EMA's CFU/mL criteria: bacterial pathogen(s) found at baseline was reduced to <10^3 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Test of cure (TOC) (Days 15-23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants | 128 | 105
Statistical Analysis 1: Comparison: Meropenem-Vaborbactam vs Piperacillin-Tazobactam; Treatment comparison of the m-MITT population; Test type: Non-Inferiority or Equivalence — The noninferiority margin was a difference of 15%. Meropenem-vaborbactam was claimed to be noninferior only if noninferiority was demonstrated for microbial eradication at TOC in the m-MITT Population; Treatment difference = 9.0, 95% CI 2-sided [-0.9 to 18.7] — Treatment difference is the estimate of the difference in the Eradication rate between the two treatment arms. The difference estimates and the 95% CIs are obtained based on Miettinen and Nurminen method

3. Primary Outcome: Proportion Of Participants In The Microbiological Evaluable (ME) Population Who Achieved A Microbiologic Outcome Of Eradication At The TOC Visit
Description: This was the primary outcome measure for the EMA. For this measure, a microbiologic outcome of Eradication was defined using the EMA's CFU/mL criteria: bacterial pathogen(s) found at baseline was reduced to <10^3 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture). The ME population included all participants who met m-MITT criteria and had a clinical outcome and microbiologic outcome at EOIVT or earlier; received <80% or >120% of expected IV doses; missed no more than 1 IV dose in the first 48 hours, missed no more than 2 consecutive IV doses; received no less than 6 doses for failure or no less than 9 doses for cure.
Time Frame: TOC (Days 15-23)
Population: ME population: all participants who met m-MITT criteria and had a clinical outcome and microbiologic outcome at EOIVT or earlier; received <80% or >120% of expected IV doses; missed no more than 1 IV dose in the first 48 hours, missed no more than 2 consecutive IV doses; received no less than 6 doses for failure or no less than 9 doses for cure.
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants | 118 | 102
Statistical Analysis 1: Comparison: Meropenem-Vaborbactam vs Piperacillin-Tazobactam; Treatment comparison of the ME population; Test type: Non-Inferiority or Equivalence — The noninferiority margin was a difference of 15%. Meropenem-vaborbactam was claimed to be noninferior only if noninferiority was demonstrated for microbial eradication at TOC in the ME Population; Treatment Difference = 5.9, 95% CI 2-sided [-4.2 to 16.0] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion Of Participants In The m-MITT Population With Overall Success
Description: This secondary outcome measure focused on the overall success in the ME population at the EOIVT and TOC visits. Overall success at TOC was defined as a clinical outcome of Cured and a microbiologic outcome of Eradication. Overall success at EOIVT was defined as a clinical outcome of Cured or Improvement and a microbiologic outcome of Eradication. Cured was defined as the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP. Improvement was defined as lessening, incomplete resolution, or no worsening of the baseline signs and symptoms of cUTI or AP, but continued IV therapy was warranted. Eradication was defined using the FDA's CFU/mL criteria that the bacterial pathogen(s) found at baseline was/were reduced to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: EOIVT (Days 5-14) and TOC (Days 15-23)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants
  EOIVT | 189 | 171
  TOC | 143 | 128

5. Secondary Outcome: Proportion Of Participants In The ME Population With Overall Success
Description: This secondary outcome measure focused on the overall success in the ME population at the EOIVT and TOC visits. Overall success was defined as a clinical outcome of Cured or Improvement and a microbiologic outcome of Eradication. Cured was defined as the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP. Improvement was defined as lessening, incomplete resolution, or no worsening of the baseline signs and symptoms of cUTI or AP, but continued IV therapy was warranted. Eradication was defined using the FDA's CFU/mL criteria that the bacterial pathogen(s) found at baseline was/were reduced to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: EOIVT (Days 5-14) and TOC (Days 15-23)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants
  EOIVT | 178 | 165
  TOC | 134 | 124

6. Secondary Outcome: Proportion Of Participants In The m-MITT Population Who Achieved A Microbiologic Outcome Of Eradication
Description: This secondary outcome measure focused on a microbiological outcome of Eradication in the m-MITT population at 5 time points: Day 3, EOIVT, end of treatment (EOT), TOC, and late follow up (LFU). Eradication was defined as a reduction in baseline bacterial pathogen(s) to <10^4 CFU/mL of urine culture (FDA) or <10^3 CFU/mL (EMA), and a negative blood culture for an organism that was identified as a uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Piperacillin-Tazobactam: Piperacillin-tazobactam (piperacillin 4 g plus tazobactam 0.5 g), infused in 100 mL normal saline, administered IV over 30 minutes, q8h, with 250 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after piperacillin-tazobactam plus saline, if clinically indicated. Treatment was administered for up to 14 days.
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants
  Day 3: FDA | 189 | 167
  EOIVT: FDA | 188 | 168
  EOT: FDA | 172 | 158
  TOC: FDA | 132 | 113
  LFU: FDA | 132 | 103
  Day 3: EMA | 186 | 164
  EOIVT: EMA | 188 | 168
  EOT: EMA | 169 | 158
  TOC: EMA | 128 | 105
  LFU: EMA | 129 | 98

7. Secondary Outcome: Proportion Of Participants In The ME Population Who Achieved A Microbiologic Outcome Of Eradication
Description: This secondary outcome measure focused on a microbiological outcome of Eradication in the ME population at 5 time points: Day 3, EOIVT, EOT, TOC, and LFU. Eradication was defined as a reduction in baseline bacterial pathogen(s) to <10^4 CFU/mL of urine culture (FDA) or <10^3 CFU/mL (EMA), and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants
  Day 3: FDA | 177 | 160
  EOIVT: FDA | 178 | 166
  EOT: FDA | 163 | 156
  TOC: FDA | 122 | 109
  LFU: FDA | 122 | 99
  Day 3: EMA | 174 | 157
  EOIVT: EMA | 178 | 166
  EOT: EMA | 160 | 156
  TOC: EMA | 118 | 102
  LFU: EMA | 120 | 94

8. Secondary Outcome: Proportion Of Participants With A Clinical Outcome Of Cure In The m-MITT Population
Description: This secondary outcome measure focused on a clinical outcome of Cure in the m-MITT Population. A clinical outcome of Cure was defined as the following: at EOIVT, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP; at EOT, TOC, and LFU, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP such that no further antimicrobial therapy was warranted. Symptom resolution did not necessarily include baseline symptoms associated with anatomic abnormalities that predisposed to cUTI, such as symptoms associated with the presence of an indwelling urinary catheter. The clinical outcome of Cure was reported only at the EOIVT, EOT, TOC, and LFU visits, and improvement was reported only at Day 3, EOIVT, and EOT visits.
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants
  Day 3: Improvement | 186 | 171
  EOIVT: Cure | 156 | 144
  EOIVT: Improvement | 33 | 30
  EOT: Cure | 179 | 167
  EOT: Improvement | 4 | 3
  TOC: Cure | 174 | 157
  LFU: Cure | 166 | 143

9. Secondary Outcome: Proportion Of Participants With A Clinical Outcome Of Cure In The Clinical Evaluable (CE) Population
Description: This secondary outcome measure focused on a clinical outcome of Cure in the CE population. A clinical outcome of Cure was defined as the following: at EOIVT, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP; at EOT, TOC, and LFU, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP such that no further antimicrobial therapy was warranted. Symptom resolution did not necessarily include baseline symptoms associated with anatomic abnormalities that predisposed to cUTI, such as symptoms associated with the presence of an indwelling urinary catheter. The clinical outcome of Cure was reported only at the EOIVT, EOT, TOC, and LFU visits, and improvement was reported only at the Day 3, EOIVT, and EOT visits.
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: CE population: all participants who received ≥1 dose of drug (MITT), had no key inclusion/exclusion criteria violations, had a clinical outcome (Cure, Improvement, Failure) at EOIVT, received 80-120% of expected IV doses, missed ≤1 IV dose in the first 48 hours, missed ≤2 consecutive IV doses overall, received ≥6 doses (Failure) or ≥9 doses (Cure).
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 248 | 258
Participants
  Day 3: Improvement | 243 | 250
  EOIVT: Cure | 202 | 206
  EOIVT: Improvement | 45 | 46
  EOT: Cure | 235 | 239
  EOT: Improvement | 7 | 6
  TOC: Cure | 231 | 224
  LFU: Cure | 220 | 209

10. Secondary Outcome: Proportion Of Participants With A Clinical Outcome Of Cure In The ME Population
Description: This secondary outcome measure focused on a clinical outcome of Cure in the ME population. A clinical outcome of Cure was defined as the following: at EOIVT, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP; at EOT, TOC, and LFU, the complete resolution or significant improvement of the baseline signs and symptoms of cUTI or AP such that no further antimicrobial therapy was warranted. Symptom resolution did not necessarily include baseline symptoms associated with anatomic abnormalities that predisposed to cUTI, such as symptoms associated with the presence of an indwelling urinary catheter. The clinical outcome of Cure was reported only at the EOIVT, EOT, TOC, and LFU visits, and improvement was reported only at the Day 3, EOIVT, and EOT visits.
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants
  Day 3: Improvement | 175 | 164
  EOIVT: Cure | 148 | 138
  EOIVT: Improvement | 30 | 30
  EOT: Cure | 170 | 161
  EOT: Improvement | 3 | 3
  TOC: Cure | 164 | 153
  LFU: Cure | 156 | 139

11. Secondary Outcome: Per-Pathogen Microbiological Outcome (FDA) In The m-MITT Population
Description: This secondary outcome measure focused on the per-pathogen (Enterobacter cloacae [E. cloacae], Enterococcus faecalis [E. faecalis], Escherichia coli [E. coli], Klebsiella pneumoniae [K. pneumoniae]) microbiological outcome of Eradication in the m-MITT population at 5 time points: Day 3, EOIVT, EOT, TOC, and LFU. Eradication was defined per the FDA criteria as a reduction in baseline bacterial pathogen(s) to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants
  Day 3: E. cloacae: number analyzed (Participants) | 10 | 5
  Day 3: E. cloacae | 10 | 3
  EOIVT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOIVT: E. cloacae | 10 | 5
  EOT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOT: E. cloacae | 10 | 5
  TOC: E. cloacae: number analyzed (Participants) | 10 | 5
  TOC: E. cloacae | 9 | 3
  LFU: E. cloacae: number analyzed (Participants) | 10 | 5
  LFU: E. cloacae | 8 | 2
  Day 3: E. faecalis: number analyzed (Participants) | 13 | 14
  Day 3: E. faecalis | 13 | 14
  EOIVT: E. faecalis: number analyzed (Participants) | 13 | 14
  EOIVT: E. faecalis | 13 | 14
  EOT: E. faecalis: number analyzed (Participants) | 13 | 14
  EOT: E. faecalis | 13 | 14
  TOC: E. faecalis: number analyzed (Participants) | 13 | 14
  TOC: E. faecalis | 7 | 12
  LFU: E. faecalis: number analyzed (Participants) | 13 | 14
  LFU: E. faecalis | 11 | 10
  Day 3: E. coli: number analyzed (Participants) | 125 | 117
  Day 3: E. coli | 124 | 106
  EOIVT: E. coli: number analyzed (Participants) | 125 | 117
  EOIVT: E. coli | 123 | 107
  EOT: E. coli: number analyzed (Participants) | 125 | 117
  EOT: E. coli | 113 | 100
  TOC: E. coli: number analyzed (Participants) | 125 | 117
  TOC: E. coli | 91 | 73
  LFU: E. coli: number analyzed (Participants) | 125 | 117
  LFU: E. coli | 91 | 69
  Day 3: K. pneumoniae: number analyzed (Participants) | 30 | 28
  Day 3: K. pneumoniae | 29 | 26
  EOIVT: K. pneumoniae: number analyzed (Participants) | 30 | 28
  EOIVT: K. pneumoniae | 29 | 26
  EOT: K. pneumoniae: number analyzed (Participants) | 30 | 28
  EOT: K. pneumoniae | 27 | 24
  TOC: K. pneumoniae: number analyzed (Participants) | 30 | 28
  TOC: K. pneumoniae | 19 | 15
  LFU: K. pneumoniae: number analyzed (Participants) | 30 | 28
  LFU: K. pneumoniae | 15 | 13

12. Secondary Outcome: Per-Pathogen Microbiological Outcome (FDA) In The ME Population
Description: This secondary outcome measure focused on the per-pathogen (E. cloacae, E. faecalis, E. coli, K. pneumoniae) microbiological outcome of Eradication in the ME population at 5 time points: Day 3, EOIVT, EOT, TOC, and LFU. Eradication was defined per the FDA criteria as a reduction in baseline bacterial pathogen(s) to <10^4 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem-Vaborbactam: Meropenem-vaborbactam (meropenem 2 grams [g] plus vaborbactam 2 g), infused in 250 milliliters (mL) normal saline, administered intravenously (IV) over 3 hours, every 8 hours (q8h), with 100 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-milligram (mg) dose every 24 hours (q24h) after a minimum of 15 doses of IV meropenem-vaborbactam plus saline, if clinically indicated. Treatment was administered for up to 14 days.
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants
  Day 3: E. cloacae: number analyzed (Participants) | 10 | 5
  Day 3: E. cloacae | 10 | 3
  EOIVT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOIVT: E. cloacae | 10 | 5
  EOT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOT: E. cloacae | 10 | 5
  TOC: E. cloacae: number analyzed (Participants) | 10 | 5
  TOC: E. cloacae | 9 | 3
  LFU: E. cloacae: number analyzed (Participants) | 10 | 5
  LFU: E. cloacae | 8 | 2
  Day 3: E. faecalis: number analyzed (Participants) | 11 | 14
  Day 3: E. faecalis | 11 | 14
  EOIVT: E. faecalis: number analyzed (Participants) | 11 | 14
  EOIVT: E. faecalis | 11 | 14
  EOT: E. faecalis: number analyzed (Participants) | 11 | 14
  EOT: E. faecalis | 11 | 13
  TOC: E. faecalis: number analyzed (Participants) | 11 | 14
  TOC: E. faecalis | 6 | 12
  LFU: E. faecalis: number analyzed (Participants) | 11 | 14
  LFU: E. faecalis | 9 | 10
  Day 3: E. coli: number analyzed (Participants) | 117 | 106
  Day 3: E. coli | 117 | 101
  EOIVT: E. coli: number analyzed (Participants) | 117 | 106
  EOIVT: E. coli | 117 | 106
  EOT: E. coli: number analyzed (Participants) | 117 | 106
  EOT: E. coli | 108 | 99
  TOC: E. coli: number analyzed (Participants) | 117 | 106
  TOC: E. coli | 84 | 71
  LFU: E. coli: number analyzed (Participants) | 117 | 106
  LFU: E. coli | 84 | 67
  Day 3: K. pneumoniae: number analyzed (Participants) | 28 | 27
  Day 3: K. pneumoniae | 28 | 25
  EOIVT: K. pneumoniae: number analyzed (Participants) | 28 | 27
  EOIVT: K. pneumoniae | 28 | 26
  EOT: K. pneumoniae: number analyzed (Participants) | 28 | 27
  EOT: K. pneumoniae | 26 | 24
  TOC: K. pneumoniae: number analyzed (Participants) | 28 | 27
  TOC: K. pneumoniae | 18 | 14
  LFU: K. pneumoniae: number analyzed (Participants) | 28 | 27
  LFU: K. pneumoniae | 15 | 12

13. Secondary Outcome: Per-Pathogen Microbiological Outcome (EMA) In The m-MITT Population
Description: This secondary outcome measure focused on the per-pathogen (E. cloacae, E. faecalis, E. coli, K. pneumoniae) microbiological outcome of Eradication in the m-MITT population at 5 time points: Day 3, EOIVT, EOT, TOC, and LFU. Eradication was defined per the EMA criteria as a reduction in baseline bacterial pathogen(s) to <10^3 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 192 | 182
Participants
  Day 3: E. cloacae: number analyzed (Participants) | 10 | 5
  Day 3: E. cloacae | 10 | 3
  EOIVT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOIVT: E. cloacae | 10 | 5
  EOT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOT: E. cloacae | 10 | 5
  TOC: E. cloacae: number analyzed (Participants) | 10 | 5
  TOC: E. cloacae | 9 | 3
  LFU: E. cloacae: number analyzed (Participants) | 10 | 5
  LFU: E. cloacae | 8 | 2
  Day 3: E. faecalis: number analyzed (Participants) | 13 | 14
  Day 3: E. faecalis | 13 | 14
  EOIVT: E. faecalis: number analyzed (Participants) | 13 | 14
  EOIVT: E. faecalis | 13 | 14
  EOT: E. faecalis: number analyzed (Participants) | 13 | 14
  EOT: E. faecalis | 12 | 13
  TOC: E. faecalis: number analyzed (Participants) | 13 | 14
  TOC: E. faecalis | 5 | 11
  LFU: E. faecalis: number analyzed (Participants) | 13 | 14
  LFU: E. faecalis | 9 | 9
  Day 3: E. coli: number analyzed (Participants) | 125 | 117
  Day 3: E. coli | 124 | 106
  EOIVT: E. coli: number analyzed (Participants) | 125 | 117
  EOIVT: E. coli | 123 | 107
  EOT: E. coli: number analyzed (Participants) | 125 | 117
  EOT: E. coli | 112 | 100
  TOC: E. coli: number analyzed (Participants) | 125 | 117
  TOC: E. coli | 89 | 68
  LFU: E. coli: number analyzed (Participants) | 125 | 117
  LFU: E. coli | 90 | 68
  Day 3: K. pneumoniae: number analyzed (Participants) | 30 | 28
  Day 3: K. pneumoniae | 29 | 24
  EOIVT: K. pneumoniae: number analyzed (Participants) | 30 | 28
  EOIVT: K. pneumoniae | 29 | 26
  EOT: K. pneumoniae: number analyzed (Participants) | 30 | 28
  EOT: K. pneumoniae | 27 | 24
  TOC: K. pneumoniae: number analyzed (Participants) | 30 | 28
  TOC: K. pneumoniae | 19 | 14
  LFU: K. pneumoniae: number analyzed (Participants) | 30 | 28
  LFU: K. pneumoniae | 15 | 12

14. Secondary Outcome: Per-Pathogen Microbiological Outcome (EMA) In The ME Population
Description: This secondary outcome measure focused on the per-pathogen (E. cloacae, E. faecalis, E. coli, K. pneumoniae) microbiological outcome of Eradication in the ME population at 5 time points: Day 3, EOIVT, EOT, TOC, and LFU. Eradication was defined per the EMA criteria as a reduction in baseline bacterial pathogen(s) to <10^3 CFU/mL of urine culture and a negative blood culture for an organism that was identified as an uropathogen (if repeated after positive at baseline blood culture).
Time Frame: Day 3, EOIVT (Days 5-14), EOT (Days 10-14), TOC (Days 15-23), and LFU (Days 22-30)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
Number analyzed (Participants) | 178 | 169
Participants
  Day 3: E. cloacae: number analyzed (Participants) | 10 | 5
  Day 3: E. cloacae | 10 | 3
  EOIVT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOIVT: E. cloacae | 10 | 5
  EOT: E. cloacae: number analyzed (Participants) | 10 | 5
  EOT: E. cloacae | 10 | 5
  TOC: E. cloacae: number analyzed (Participants) | 10 | 5
  TOC: E. cloacae | 9 | 3
  LFU: E. cloacae: number analyzed (Participants) | 10 | 5
  LFU: E. cloacae | 8 | 2
  Day 3: E. faecalis: number analyzed (Participants) | 11 | 14
  Day 3: E. faecalis | 11 | 14
  EOIVT: E. faecalis: number analyzed (Participants) | 11 | 14
  EOIVT: E. faecalis | 11 | 14
  EOT: E. faecalis: number analyzed (Participants) | 11 | 14
  EOT: E. faecalis | 10 | 13
  TOC: E. faecalis: number analyzed (Participants) | 11 | 14
  TOC: E. faecalis | 4 | 11
  LFU: E. faecalis: number analyzed (Participants) | 11 | 14
  LFU: E. faecalis | 8 | 9
  Day 3: E. coli: number analyzed (Participants) | 117 | 106
  Day 3: E. coli | 117 | 101
  EOIVT: E. coli: number analyzed (Participants) | 117 | 106
  EOIVT: E. coli | 117 | 106
  EOT: E. coli: number analyzed (Participants) | 117 | 106
  EOT: E. coli | 107 | 99
  TOC: E. coli: number analyzed (Participants) | 117 | 106
  TOC: E. coli | 82 | 67
  LFU: E. coli: number analyzed (Participants) | 117 | 106
  LFU: E. coli | 83 | 66
  Day 3: K. pneumoniae: number analyzed (Participants) | 28 | 27
  Day 3: K. pneumoniae | 28 | 23
  EOIVT: K. pneumoniae: number analyzed (Participants) | 28 | 27
  EOIVT: K. pneumoniae | 28 | 26
  EOT: K. pneumoniae: number analyzed (Participants) | 28 | 27
  EOT: K. pneumoniae | 26 | 24
  TOC: K. pneumoniae: number analyzed (Participants) | 28 | 27
  TOC: K. pneumoniae | 18 | 13
  LFU: K. pneumoniae: number analyzed (Participants) | 28 | 27
  LFU: K. pneumoniae | 15 | 11

15. Secondary Outcome: Pharmacokinetic (PK) Characterization Of Plasma Exposure Of Meropenem/Vaborbactam
Description: This outcome measure focused on PK assessment of participants in the meropenem/vaborbactam group who met MITT criteria and had at least 1 plasma PK sample drawn. Sparse PK sampling on Day 1 was performed 3-3.5 hours and 5-6 hours after the start of the first 3-h IV study drug infusion. Samples were not collected around the 30-minute infusions. Samples were collected from both groups to maintain the blind; however, only PK samples for the meropenem/vaborbactam group were analyzed. The area under the curve (AUC) was generated using a Population PK model and post hoc estimates of each participants' PK parameters, including AUC0-24, were generated.
  The AUC during 24 hours (AUC0-24) for Day 1 and at steady-state are presented in micrograms (ug)·hour/mL.
Time Frame: Day 1
Population: PK population: Participants in the MITT population (all participants screened, randomized, and received at least 1 dose of study drug) and had at least 1 plasma PK sample drawn. Due to renal impairment, 28 participants received a reduced dose of the study drug (1 g meropenem/1 g vaborbactam).
Measure: Mean (Standard Deviation); unit: ug·hour/mL
Groups:
- Meropenem-Vaborbactam: Meropenem-vaborbactam (meropenem 2 g plus vaborbactam 2 g), infused in 250 mL normal saline, administered IV over 3 hours, q8h, with 100 mL saline administered over 30 minutes q8h. Levofloxacin tablets administered orally as a 500-mg dose q24h after a minimum of 15 doses of IV meropenem-vaborbactam plus saline, if clinically indicated. Treatment was administered for up to 14 days.
  AUC0-24 Steady-State estimates not available for 2 participants who received >3 doses.
Arm/Group | Meropenem-Vaborbactam
Number analyzed (Participants) | 272
ug·hour/mL
  AUC0-24: Day 1 | 803 (45.3)
  AUC0-24: Steady-State | 798 (60.6)

ADVERSE EVENTS:
Time Frame: Days 1 (Screening) through 30 (Follow Up).
Arm/Group | Meropenem-Vaborbactam | Piperacillin-Tazobactam
All-Cause Mortality (participants affected / at risk) | 2/272 | 2/273
Serious Adverse Events (participants affected / at risk) | 11/272 | 12/273
Other Adverse Events (participants affected / at risk) | 36/272 | 31/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Meropenem-Vaborbactam (N=272) | Piperacillin-Tazobactam (N=273)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Salpingo-oophoritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Meropenem-Vaborbactam (N=272) | Piperacillin-Tazobactam (N=273)
Headache (Nervous system disorders) | 24 | 12
Diarrhoea (Gastrointestinal disorders) | 9 | 12
Infusion Site Phlebitis (General disorders) | 6 | 2
Vaginal Infection (Infections and infestations) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No